CONTRACT RESEARCH ORGANIZATION: SPONSOR:

AMS Advanced Medical Services GmbH DS Biopharma

Am Exerzierplatz 2 Trintech Building

D-68167 Mannheim South County Business Park

Phone: +49 (0)621 / 70095 100 Leopardstown

Fax: +49 (0)621 / 70095 140 Dublin 18,

Republic of Ireland

# **Statistical Analysis Plan**

### for Clinical Trial Protocol DS107G-05-AD3

Study Title A Randomised, Double-blind, Placebo-controlled Study to Assess

the Efficacy and Safety of Orally Administered DS107 in Adult

Patients with Moderate to Severe Atopic Dermatitis

**Study Medication** DS107 Capsules

**Type of Study** Multicenter, double-blind, placebo controlled, 2-arm, Phase II

study with 16 weeks of active treatment and a 4 week follow up

period

Objectives of Study The primary objective is to compare the efficacy of orally

administered DS107 versus placebo, in the treatment of adult

patients with moderate to severe Atopic Dermatitis (AD).

The secondary objective is to assess the safety of orally administered DS107 versus placebo, in adult patients with

moderate to severe AD.

**Sponsor Study No.** DS107G-05-AD3

**EudraCT-No.:** 2019-000932-25

AMS Study No. DS23349

**Responsible** Florian Schelz

Biometrician AMS Advanced Medical Services GmbH

**Author** Florian Schelz

AMS Advanced Medical Services GmbH

**Date** Sep 24, 2020

**Status of Document** Final Version 1.0

Pages 34

CONFIDENTIAL

## Change management

| Version | Date | Author | Description of changes |
|---|---|---|---|
| 0.1 | May 19, 2020 | Florian Schelz | First Draft Version |
| 0.2 | Sep 07, 2020 | Florian Schelz | Second draft Version after Sponsor Review |
| 0.3 | Sep 21, 2020 | Florian Schelz | Third draft Version after second Sponsor |
| | | | Review |
| 1.0 | Sep 24, 2020 | Florian Schelz | Final Version |

# **Table of Contents**

| Table of C | Contents | 3 |
|---|---|---|
| List of Ab | obreviations and Definition of Terms | 5 |
| 1 | Introduction | 7 |
| 1.1 | Study Objectives | 7 |
| 1.2 | General Study Design | 7 |
| 1.3 | Study Population | 7 |
| 1.4 | Study Medication | 8 |
| 1.5 | Randomisation | 8 |
| 1.6 | Interim Analysis | 8 |
| 1.7 | Time Schedule / Study Duration | 9 |
| 2 | Sample Size | 9 |
| 3 | Analysis Populations | 10 |
| 4 | Data Handling | 11 |
| 4.1<br>4.1.1<br>4.1.2<br>4.1.3<br>4.1.4<br>4.1.5 | General Data sources Coding Visits Baseline value Missing values | 11<br>11<br>11<br>11<br>11 |
| 4.2<br>4.2.1<br>4.2.2<br>4.2.3<br>4.2.4<br>4.2.5<br>4.2.6<br>4.2.7<br>4.2.8<br>4.2.9<br>4.2.10<br>4.2.11<br>4.2.12<br>4.2.13 | Algorithms for data calculations and modifications Study Day Age BMI Validated Investigator Global Assessment (vIGA-AD <sup>TM</sup> ) Eczema Area Severity Index (EASI) Pruritus NRS Body Surface Area (BSA) Dermatology Life Quality Index (DLQI) Questionnaire Patient Orientated Eczema Measure (POEM) SCORing Atopic Dermatitis (SCORAD) Athens Insomnia Scale (AIS) Patient Oriented SCORAD (PO-SCORAD) Study medication: Intake and duration of intake | 12<br>12<br>12<br>12<br>12<br>12<br>13<br>13<br>13<br>13<br>14<br>14<br>14 |

## Statistical Analysis Plan DS107G-05-AD3 Version 1.0 (final), 24-Sep-2020

| 4.2.14<br>4.2.15 | Previous vs. concomitant medication<br>Adverse events | 15<br>15 |
|---|---|---|
| 5 | Blind Data Review Meeting | 15 |
| 6 | General Methodology | 16 |
| 6.1 | Primary Endpoint Evaluation | 16 |
| 6.2 | Descriptive, Exploratory Analyses | 16 |
| 6.3 | Subgroup analyses | 17 |
| 7 | Final analysis | 17 |
| 7.1 | Demographic and other baseline characteristics | 17 |
| 7.2 | Efficacy - Primary Endpoint Evaluation | 17 |
| 7.3 | Efficacy - Secondary Endpoints Evaluation | 17 |
| 7.4 | Efficacy - Exploratory Endpoints Evaluation | 19 |
| 7.5 | Safety Evaluation | 20 |
| 7.6 | Further Analyses | 22 |
| 8 | Tables and Figures | 23 |
| 9 | References | 34 |

### List of Abbreviations and Definition of Terms

AD Atopic Dermatitis

AE Adverse Event

AIS Athens Insomnia Scale

AMS Advanced Medical Services GmbH

ATC Anatomical Therapeutic Chemical

BDRM Blind Data Review Meeting

BMI Body Mass Index

BSA Body Surface Area

DGLA Dihomo-Gamma-Linolenic Acid

DLQI Dermatology Life Quality Index

EASI Eczema Area and Severity Index

ECG Electrocardiography

eCRF electronic Case Report Form

FAS Full Analysis Set

g Gram

GLMM Generalised Linear Mixed Model

ICH International Conference on Harmonization

IGA Investigator Global Assessment

IMP Investigational Medicinal Product

IWRS Interactive Web Response System

kg Kilogram

MAR Missing at Random

MedDRA Medical dictionary for Drug Regulatory Affairs

MMRM Mixed Model with Repeated Measures

NRS Numeric Rating Scale

No. Number

POEM Patient Orientated Eczema Measure

PO-SCORAD Patient Oriented Scoring of Atopic Dermatitis

PPS Per-Protocol Set

SAE Serious Adverse Event

SAP Statistical Analysis Plan

SAS Statistical Analysis System

SCORAD Scoring of Atopic Dermatitis

SOC System Organ Class

SOP Standard Operating Procedure

TMF Trial Master File

vIGA-AD<sup>TM</sup> Validated Investigator Global Assessment Scale for Atopic Dermatitis

WHO World Health Organisation

#### 1 Introduction

This Statistical Analysis Plan (SAP) refers to the Trial Protocol DS107G-05-AD3, final version 5.0 (EU) and version 5.1 (US) dated March 18, 2020 which includes the previously approved versions of the protocol. The SAP will be finalised before any analysis will be conducted. The specifications included in this SAP which have not been mentioned in the study protocol, are restricted to statistical issues, and have no impact on the clinical conduct of the trial.

This SAP describes the analysis to be performed at the end of the trial.

Additions or changes to the analysis planned in this SAP may be defined during the BDRM (Blind Data Review Meeting) and documented in the BDRM protocol which will be approved by the BDRM participants.

The document is written in compliance with the ICH Guidelines E9 and the *AMS* SOP ST-02.01 (Statistical Analysis Plan).

### 1.1 Study Objectives

The primary objective of this clinical trial is to compare the efficacy of orally administered DS107 (2g) versus placebo, in the treatment of adult patients with moderate to severe AD. The secondary objective is to assess the safety of orally administered DS107 (2g) versus placebo, in adult patients with moderate to severe AD.

It is planned to test the trial medication versus placebo in a total of 220 patients.

## 1.2 General Study Design

This clinical trial will be carried out as a randomised, placebo-controlled, double-blind, parallel group, multi-centre 2-arm Phase 2 study to investigate the efficacy of orally administered DS107 in AD patients.

It is planned that at least 220 patients suffering from moderate to severe AD will be included in this study. All patients will sign an informed consent and undergo screening for study eligibility.

Before the comparative treatment period can commence, patients will return to the site for a baseline assessment of their disease and eligible patients will be randomly allocated to one of the treatment regimens in a 1:1 randomization:

- 2g DS107 (4 DS107 capsules) orally administered once daily for 16 weeks
- Placebo (4 placebo capsules) orally administered once daily for 16 weeks

There is a 4 week follow-up period.

To maintain the double-blind conditions, DS107 capsules and placebo will be identical in appearance.

#### 1.3 Study Population

The study population will consist of male and female patients with confirmed diagnosis of AD aged 18 years or older.

### 1.4 Study Medication

The following medication supplies will be used in the study:

### DS107 capsules:

Each DS107 capsule contains 500mg DGLA as an active ingredient in an opaque, oval soft gelatin capsule.

#### Placebo capsule:

Each matching placebo capsule contains 500mg of liquid paraffin in an opaque oval soft gelatin capsule.

#### 1.5 Randomisation

Approximately 220 patients will be randomized into double-blind treatment groups in a 1:1 ratio by an IWRS.

- 2g DS107 (4 DS107 capsules) administered once-daily for 16 weeks
- Placebo (4 placebo capsules) orally administered once-daily for 16 weeks

A randomization list permuted by blocks and stratified by site will be generated by the Sponsor or its designee. The randomization schedule with study drug assignments will be generated prior to the start of the study and will be known only to the individuals responsible for labelling the study drug, the statisticians generating the schedule and the IWRS team responsible for implementing the schedule. The IWRS will assign a medication kit number to each patient and the contents will be based on the randomization code.

At the investigational site, each patient will be assigned a patient identifier number during screening that will be used on all patient documentation. The patient identifier number will contain the site number and the patient number assigned in numerical order at the Screening Visit (e.g.: 102-10 for the tenth patient screened at the site number 02). Patient numbers will be assigned in ascending order starting with 01.

The treatment assignment procedure will use blocks of sufficient size to maintain a blind and balance across treatment arms. Following successful completion of the screening/baseline evaluations and confirmation that the patient is eligible for participation, the patient will be randomised to treatment. This will be performed by the Investigator using the IWRS which will assign a medication number to the patient.

### 1.6 Interim Analysis

An interim analysis may be conducted after at least 50% of planned enrolled patients have completed their Week 16 assessments or an early termination visit. The interim analysis will be conducted in accordance with sponsor standard operating procedure (SOP) "Interim Analysis of Clinical Studies".

An unblinded interim analysis will be performed by an unblinded independent statistician. Interim data and the results of interim analyses will not be accessible by anyone other than the unblinded statistician. The sponsor will remain blinded with procedures in place to ensure the confidentiality of the interim data, as per the sponsor SOP "Interim Analysis of Clinical Studies".

The unblinded statistician will make one of the following recommendations to the sponsor based solely upon the primary efficacy endpoints:

- Modify the sample size
- Continue the study as originally planned
- Stop the study due to futility

Further details will be described in an interim statistical analysis plan. No  $\alpha$  adjustment will be executed.

Due to the rapidly evolving COVID-19 situation at both a global and country level, a modification to the prospectively planned sample size may be necessary if patient recruitment is not feasible and must be stopped. The interim analysis will safeguard the integrity of the trial and inform whether further patient recruitment is required when conditions at participating sites are amenable to re-initiation of patient recruitment.

### 1.7 Time Schedule / Study Duration

Patients will come to the clinic on 8 occasions: at Screening/Visit 1, Baseline/Visit 2, Week 4/Visit 4, Week 8/Visit 5, Week 12/Visit 6, Week 16/Visit 7 (end of treatment), Week 18/ Visit 8 (follow up) and Week 20/Visit 9 (follow-up). A telephone visit will also be performed at Week 1/Visit 3.

Patients who discontinue the study early will be asked to attend the investigative site as soon as possible so that assessments scheduled for Visit 7 can be conducted at an Early Termination visit.

In the event that treatment is occurring, a wash out period of up to 4 weeks may be necessary. At the Screening Visit, after giving informed consent to participate, patients will be assessed using the screening examinations. Eligible patients with confirmed AD using the American Academy of Dermatology Consensus Criteria and who meet all the inclusion criteria and do not meet the exclusion criteria at the baseline visit will be enrolled.

During the treatment period and follow-up period patients will be restricted from using any other treatment for AD, with the exception of the same emollients they have been consistently using since the screening visit.

## 2 Sample Size

In the Phase 2a trial, IGA response rates of 21.6% and 11.8% were observed for DS107 and placebo respectively resulting in a difference in response rates of 9.8%. Due to the prolonged treatment period of 16 weeks, a clinically relevant difference in IGA response rates of 15% was expected for the current study.

Assuming a placebo response rate of 12% and a true response rate difference of 15% at Week 16 and using a two-sided Chi-Square test on a significance of 5%, then 220 evaluable patients (110 patients per treatment arm) will be needed for 80% power to detect this difference as statistically significant. As the following table shows, the number of patients needed for the discovery of a 15% response rate difference depends also on the placebo response rate shown in the left column of the table as decimal numbers:

Number of patients per study group required under the assumptions as follows
Chi-square test, 2 x 2 table, Two Proportions, two-sided.
Sample Size 1 as a function of H1: Proportion 1 and Power.
H1: Proportion 2 - Proportion 1=0,15 Significance Level=0,05 Sample Size 2 / Sample Size 1=1

| H1: Proportion 1 | | Power | |
|----------------------------|-------|-------|-------|
| = Response Rate<br>Placebo | 0,7 | 0,8 | 0,9 |
| 0,06 | 63,4 | 80,3 | 107,0 |
| 0,08 | 71,2 | 90,2 | 120,3 |
| 0,10 | 78,6 | 99,6 | 132,8 |
| 0,12 | 85,5 | 108,4 | 144,6 |
| 0,14 | 92,0 | 116,6 | 155,6 |
| 0,16 | 98,0 | 124,3 | 165,9 |
| 0,18 | 103,6 | 131,4 | 175,4 |
| 0,20 | 108,8 | 138,0 | 184,2 |

It was assumed that similar estimations apply to the primary endpoint EASI-75.

### 3 Analysis Populations

The assignment of individual patients to the analysis sets will be determined by the members of the BDRM. The patients will be assigned to the following analysis sets before unblinding:

- 1. Enrolled Set: The Enrolled Set consists of all patients who sign informed consent.
- 2. Screen Failures: Screen Failures are patients from the Enrolled Set who do not meet the eligibility requirements and are withdrawn from the study prior to randomisation.
- 3. Randomised Set: The Randomised Set consists of all patients who are randomised to the study.
- 4. Safety Analysis Set (SAS): The Safety Analysis Set (SAS) consists of all patients who received at least one dose of the medication. SAS is the analysis population for all safety endpoints. Analysis will be done according to the actual treatment patients received.
- 5. Full Analysis Set (FAS): The Full Analysis Set (FAS) consists of all patients who were randomised to the study and received at least one dose of study medication. FAS is the primary analysis population for efficacy endpoints. Analysis will be done according to the treatment patients were randomised to.
- 6. Per-Protocol Set (PPS): The Per Protocol Set (PPS) is the subset of FAS who completed the study without any major violations. Protocol violations will be assessed for each patient in a blinded fashion prior to database lock at a Blind Data Review Meeting (BDRM), and the PPS will also be finalised during this meeting. PPS is a supportive analysis population for efficacy endpoints. Analysis will be done according to the treatment patients were randomised to.

For PPS the primary endpoint will only be evaluated in an exploratory sense.

### 4 Data Handling

#### 4.1 General

#### 4.1.1 Data sources

Most of the data collected in connection with this trial are recorded in an eCRF (electronic Case Report Form). The diary data (NRS, AIS, IMP compliance etc) is recorded in the IRT system. All patient data will be entered by the investigator. Details can be found in the data handling manual for this study. The entered data are subjected to plausibility checks. These are detailed in the data validation plan for this study.

### **4.1.2 Coding**

The process of coding is performed according to the *AMS* internal Coding SOP and relevant Coding guidelines (e.g. 'MedDRA Points to consider' / 'Best Practices for the use of the WHO Drug Dictionaries').

The data to be coded is extracted into a coding database where the coding is performed. Details of the coding database, the items to be coded, the frequency of coding and the 'MedDRA' version used for coding of diseases and adverse events and the WHO DD version used for coding of medications and the update frequency of the dictionaries are defined in the Coding Specification.

#### **4.1.3** Visits

The analysis visits and points in time will be presented as documented in the database.

#### 4.1.4 Baseline value

The last non-missing value prior to first treatment will be referred to as baseline value and will be used for change from baseline calculations.

#### 4.1.5 Missing values

If only the day is not known completely, for onset dates or start dates missing day information will be assumed as the 1<sup>st</sup>. If both day and month are missing, the 1<sup>st</sup> January will be used. For stop dates missing day information will be imputed as the last of the month, if both day and month are missing, the 31<sup>st</sup> December will be used.

However, if for AEs it is not clear whether the event started prior to or in the treatment period, the onset at day of first treatment will be assumed.

If it is not clear due to a missing or incomplete stop date of a medication whether the medication was taken at least once after the first treatment of the patient, a stop date after the day of the first patient visit will be assumed. The medication will therefore be classified as "concomitant medication". If it is not clear due to a missing or incomplete start date of a medication whether the medication was taken at least once before the first treatment of the patient, a start date before the day of the first patient visit will be assumed. The medication will therefore be classified as "previous medication" (cf. section 4.2.14).

Data from patients who prematurely terminate the trial will be used to the maximum extent possible.

The primary statistical analysis assumes "Missing At Random (MAR)" when handling missing data. The treatment effect obtained under the MAR assumption is essentially that which could have been reached if all patients had fully adhered to treatment or, in other words, the effect a patient may expect if they take the medication as directed. This is sometimes known as the 'de jure' or 'efficacy' estimand. Due to the lack of perfect adherence in practice, the 'de facto' or effectiveness treatment effect will also be estimated. This estimand includes assumptions regarding the treatment effects that could be expected to occur when patients discontinue treatment. The jump to reference method described by Carpenter et al. (2013) will be used to estimate the de facto estimand, using the placebo arm as the reference. This is based on the assumption that patients who discontinue from study drug have no alternative oral treatment option suitable for longer-term use and so their responses are likely to revert to those of the placebo group. An additional sensitivity analysis will evaluate patients who received rescue medication as treatment failures from the visit onwards where rescue treatment started. The sensitivity analyses for missing data will be performed on the FAS only.

### 4.2 Algorithms for data calculations and modifications

### 4.2.1 Study Day

The Study Day of an assessment or event will be defined as

Study Day = Date of Assessment - Date of first treatment +1

for assessments performed at/after date of first treatment.

For assessments prior date of first treatment the definition is as follows:

Study Day = Date of Assessment - Date of first treatment

For patients without treatment, study day will not be calculated.

### 4.2.2 Age

The age of patients at time of consent [in years] is used as documented in the eCRF.

#### 4.2.3 BMI

The Body Mass Index (BMI) of patients at screening is used as documented in the eCRF.

# 4.2.4 Validated Investigator Global Assessment (vIGA-AD<sup>TM</sup>)

The clinical severity of AD will be evaluated by the Investigator at each visit using the vIGA-AD<sup>TM</sup> scale.

The vIGA-AD<sup>TM</sup> scale awards a score of 0-4 based on a 5-point severity scale from clear to severe disease (0 = clear, 1 = almost clear, 2 = mild disease, 3 = moderate disease, 4 = severe disease). The scale uses clinical characteristics of erythema, infiltration, papulation and oozing/crusting as scoring guidelines for the overall severity assessment. vIGA-AD<sup>TM</sup> will be assessed at every clinic visit.

### 4.2.5 Eczema Area Severity Index (EASI)

EASI quantifies the severity of a patient's AD based on both lesion severity and the percent of BSA affected (Hanifin et al. 2001). The EASI is a composite score ranging from 0-72 that takes

into account the degree of erythema, induration/papulation, excoriation, and lichenification (each scored from 0 to 3 separately, half points are permitted) for each of four body regions, with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body.

#### 4.2.6 Pruritus NRS

Severity of pruritus related to AD will be self-assessed by patients daily using the NRS. Patients will be asked to estimate the intensity of pruritus at its worst over the previous 24 hours. The Pruritus NRS is a single-question assessment tool that will be used to assess the patient's worst itch as a result of AD in the previous 24 hours. Patients will score their pruritus due to AD on a scale of 0 - 10, with 0 (no itch) and 10 (worst itch imaginable) (Phan et al. 2012). Patients will complete the rating scale daily starting at screening through to the last study visit.

The baseline NRS is defined as the prorated average of the NRSs reported continuously for 7 days right before and on the baseline visit (i.e. study day -6 to day 1). For post-baseline NRS, the mean weekly worst itch NRS is calculated as the prorated average of the reported daily NRS within the week. For example, if there are 3 scores in a week, the prorated average = (score1 + score2 + score3)/3.

### 4.2.7 Body Surface Area (BSA)

The overall BSA affected by AD will be evaluated (from 0 to 100%) at each visit. One patient's palm represents 1% of his/her total BSA. BSA will be evaluated at every clinic visit.

### 4.2.8 Dermatology Life Quality Index (DLQI) Questionnaire

The effect of AD on patient quality of life will be self-assessed by the patient at every clinic visit starting from baseline, using the DLQI developed by Finlay and Khan (1994).

DLQI has a maximum value of thirty based on the patients response to ten questions scored according to the following scale:

- Very Much = 3
- A lot = 2
- A little = 1
- Not at all = 0
- Not relevant = 0
- Question unanswered = 0
- Question 7: "prevented work or studying" = 3

### **4.2.9** Patient Orientated Eczema Measure (POEM)

The POEM will be assessed at each clinic visit, except the screening visit. The POEM developed by Charman et.al. 2004 is a self-assessment of disease severity by the patient. POEM has a maximum value of twenty eight based on the patient's response to seven questions scored according to the following scale:

• No Days = 0

- 1-2 Days = 1
- 3-4 Days = 2
- 5-6 Days = 3
- Everyday = 4

## **4.2.10 SCORing Atopic Dermatitis (SCORAD)**

SCORAD will be measured at each clinic visit, except the screening visit. The SCORAD grading system was developed by the European Task Force on Atopic Dermatitis (1993) and has been a standard tool to assess the AD severity in clinical studies. Six items (erythema, edema/papulation, oozing/crusts, excoriation, lichenification, and dryness) will be selected to evaluate the AD severity. The overall BSA affected by AD will be evaluated (from 0 to 100%) and included in the SCORAD scores. Loss of sleep and pruritus will be evaluated by patients on a visual analog scale (0-10). The sum of these measures represents the SCORAD which can vary from 0 to 103.

### 4.2.11 Athens Insomnia Scale (AIS)

The severity of sleep disturbance will be self-assessed daily starting from baseline using the Athens Insomnia Scale (AIS).

The AIS is a self-administered psychometric instrument consisting of eight items. The first five items of the AIS (assessing difficulty with sleep induction, awakenings during the night, early morning awakening, total sleep time, and overall quality of sleep) correspond to Criterion A for the diagnosis of insomnia according to ICD-10 (International Statistical Classification of Diseases and Related Health Problems 10<sup>th</sup> Revision), while the requirements of a minimum frequency (at least three times a week) and duration (1 month) of any complaint correspond to Criterion B of the ICD-10. The ICD-10 requirements of marked distress caused by the sleep problem and/or interference with ordinary activities of daily living (Criterion C) are covered through the strictly subjective nature of the response options for every item of the scale as well as through the content of the last three items pertaining to the next day consequences of insomnia (problems with sense of well-being, functioning, and sleepiness during the day).

Each item of the AIS can be rated 0-3.

The responders are requested to rate positively if they had experienced the sleep difficulty described in each item at least three times a week between the study visits (Soldatos et al. 2000).

The baseline AIS is defined as the prorated average of the AISs reported continuously for 7 days right before and on the baseline visit (i.e. study day -6 to day 1). For post-baseline AIS, the mean weekly worst itch AIS is calculated as the prorated average of the reported daily AIS within the week. For example, if there are 3 scores in a week, the prorated average = (score1 + score2 + score3)/3.

## **4.2.12 Patient Oriented SCORAD (PO-SCORAD)**

The PO-SCORAD will be measured at each clinic visit, except the screening visit. The PO-SCORAD is the SCORAD completed by the patients themselves. It is a self-evaluation tool developed by the European Task Force on Atopic Dermatitis (2011). Six items (erythema, edema/papulation, oozing/crusts, excoriation, lichenification, and dryness) will be selected to evaluate the AD severity. The overall surface affected, loss of sleep and pruritus will also be evaluated by patients on a visual analog scale.

### 4.2.13 Study medication: Intake and duration of intake

The duration of intake of study medication will be calculated as day of last dispensed of study medication minus day of first dispensed of study medication plus one.

The intake of study medication will be calculated as the number of capsules dispense per visit.

#### 4.2.14 Previous vs. concomitant medication

Previous medications are those medications taken at least once before the first treatment of the patient. Concomitant medications are those medications taken at least once at/after the first treatment of the patient.

#### 4.2.15 Adverse events

AEs with onset during or after administration of first study medication (study day 1) are defined as treatment emergent.

### 5 Blind Data Review Meeting

A BDRM will be held prior to database hard lock/unblinding where **AMS** and Sponsor representatives will assess protocol deviations as major or minor with regard to their influence on any of the analysis variables and to determine patient inclusion in the analysis sets.

The **AMS** biostatistician will prepare blinded review listings. Deviations not apparent in the clinical database (e.g. findings during monitoring of the investigational site) will be contributed by the sponsor's clinical project leader.

The decisions of the BDRM will be documented in writing and will be approved by signature of the attendees and may potentially amend methodology/analysis set definitions planned in this SAP.

The discussion in the review meeting will include but may not be restricted to the following topics:

- Violations of the study protocol including violations of inclusion/exclusion criteria
- Identification of patients randomised but not treated
- Impact assessment of prohibited medications
- Patients without efficacy data
- Patients where blind was broken prior to formal unblinding of the study
- Procedural deviations at the trial sites which are not reflected in the clinical database
- Premature patient discontinuations (reason and timing).
- Patients with COVID-19
- Patients with Week 16 visit window violations
- Assessment of impact of the COVID19 pandemic on visits occurring during COVID19 pandemic vs. other visits

Full details on the reviews performed and the decisions made in the BDRM will be given in the BDRM protocol.

## 6 General Methodology

All analyses will be performed using SAS Version 9.4 or higher.

If not mentioned otherwise analyses will be stratified by treatment group displaying the following treatment groups (in this ordering): DS107, Placebo, Total. Therefore treatment will not be mentioned explicitly as stratification variable usually.

All eCRF data will be listed, therefore listings may not be mentioned explicitly.

In listings the patient's screening number will be used as the main patient identifier. Usually listings will be sorted by treatment, patient's screening number and (if applicable) visit/point in time.

### 6.1 Primary Endpoint Evaluation

The primary endpoint variables will be:

- the proportion of patients achieving an vIGA-AD<sup>TM</sup> score of 0 (clear) or 1 (almost clear) and a decrease of at least 2 points in vIGA-AD<sup>TM</sup> from baseline to Week 16.
- the proportion of patients achieving EASI-75 (≥75% improvement from baseline) at Week 16.

Both primary endpoints will be analysed using a Generalised Linear Mixed Model (GLMM) with treatment arm, visit, their interaction treatment-by-visit, and baseline vIGA-AD<sup>TM</sup> value as factors, and with patient as random effect; this model will especially be used to estimate missing data and the treatment effects at Week 16 taking missing data into account. The primary analysis will be based on the FAS, and repeated for the PPS as a supportive sensitivity analysis. Success in either of the primary endpoints denotes successful proof of efficacy.

If rescue medication is used, the patient will be specified as a non-responder from the time the rescue is used.

The handling of missing data in regards with primary statistical analysis and further sensitivity analysis using the jump to reference method to estimate the de facto estimand and analysing patients who received rescue medication as treatment failures are described in section 4.1.5.

## **6.2** Descriptive, Exploratory Analyses

Categorical variables will be displayed by absolute and relative frequencies (percentages). Percentages for categorical variables will be based on all non-missing values (=100%). Percentages will be rounded to one decimal place and therefore, there may be occasions when the total of the percentages does not exactly equal 100%.

Continuous variables will be summarised with number of observations, mean, standard deviation, median, minimum, maximum and the 5%, 25%, 75% and 95% quantiles. These descriptive statistics will be calculated for absolute values and for absolute differences to baseline, where appropriate.

### 6.3 Subgroup analyses

The primary endpoint will be conducted also by subgroups. The following subgroups will be considered:

• Baseline IGA (3, 4)

Further subgroups may be defined in the BDRM protocol if reasonable.

### 7 Final analysis

The following chapter summarises all analyses planned for the analysis of data collected within this trial.

### 7.1 Demographic and other baseline characteristics

Analyses of demographic will be performed as described in chapter 6.2 with the Randomised Set, details of the used analysis sets are described in chapter 8. The analysis will only be displayed overall. The following variables will be analysed:

- Age at time of consent [years]
- Gender (male, female)
- Height [cm]
- Weight [kg]
- BMI  $[kg/m^2]$
- Race (American Indian or Alaska Native, Asian, Black or African American, Native Hawaiian or Other Pacific Islander, White, Other)
- Ethnicity (Hispanic or Latino, Not Hispanic or Latino)

Demographic data will be listed.

The incidence of previous and concomitant diseases ("Medical History") will be displayed by MedDRA primary System Organ Class (SOC) and Preferred Term for the FAS.

## 7.2 Efficacy - Primary Endpoint Evaluation

Descriptive statistics will be provided for the two primary endpoints separately with the FAS.

Both primary efficacy endpoints will be analysed as defined in chapter 6.1 with the FAS.

These analyses will be displayed not only overall but also by subgroups as defined in chapter 6.3. The overall analysis will be repeated in an exploratory sense with the PPS.

## 7.3 Efficacy - Secondary Endpoints Evaluation

All secondary efficacy analyses will be performed as described in chapter 6.2 with the FAS only.

IGA and EASI-75 responders at other time points will also be analysed using a GLMM model similar to that described in Section 6.1.

The efficacy variables and their changes from baseline will be summarized with descriptive statistics per treatment group and visit. This applies to the vIGA-AD<sup>TM</sup>, EASI, NRS scores for

pruritus, DLQI, POEM, SCORAD, AIS and PO-SCORAD. Change from baseline endpoints will be analysed using Mixed Model with Repeated Measures (MMRM) with Treatment Arm, Visit and Treatment x Visit Interaction as a factors and baseline value as a covariate, to account for missing data. For vIGA-AD<sup>TM</sup> as a 5-level ordinal variable, mixed ordinal logistic regression will be used with factors defined as above and IGA at baseline as a factor too.

If rescue medication is used, the patient will be specified as a non-responder from the time the rescue is used.

The following parameters will be analysed as described above:

- Proportion of patients achieving a vIGA-AD<sup>TM</sup> score of 0 (clear) or 1 (almost clear) and a
  decrease of at least 2 points in vIGA-AD<sup>TM</sup> in treated population compared to placebo
  population from baseline to Week 4, 8, 12, 18 and 20
- Change in proportion of patients achieving a vIGA-AD<sup>TM</sup> score of 0 (clear) or 1 (almost clear) and a decrease of at least 2 points in vIGA-AD<sup>TM</sup> in treated population compared to placebo population from Week 16 to Week 18 and 20.
- Absolute proportion of patients achieving EASI-75 (≥75% improvement from baseline) in treated population compared to placebo population at Week 4, 8, 12, 18 and 20
- Change from baseline in vIGA-AD<sup>TM</sup> score in treated population compared to placebo population to Week 4, 8, 12, 16, 18 and 20
- Change from Week 16 in vIGA-AD<sup>TM</sup> score in treated population compared to placebo population to Week 18 and 20.
- Change from baseline in EASI in treated population compared to placebo population to Week 4, 8, 12, 16, 18 and 20
- Change from Week 16 in EASI in treated population compared to placebo population to Week 18 and 20.
- Absolute proportion of patients achieving a decrease of at least 4 points in worst itch NRS in treated population compared to placebo population from baseline to Week 4, 8, 12, 16, 18 and 20. The NRS endpoint should be recorded weekly (descriptive values), as defined in section 4.2.6 and p-values only provided for the weeks defined in the endpoint.
- Absolute proportion of patients achieving a decrease of at least 3 points in worst itch NRS in treated population compared to placebo population from baseline to Week 4, 8, 12, 16, 18 and 20. The NRS endpoint should be recorded weekly (descriptive values), as defined in section 4.2.6 and p-values only provided for the weeks defined in the endpoint.
- Change from baseline in worst itch NRS in treated population compared to placebo population to Week 4, 8, 12, 16, 18 and 20. The NRS endpoint should be recorded weekly (descriptive values), as defined in section 4.2.6 and p-values only provided for the weeks defined in the endpoint.
- Change from Week 16 in worst itch NRS in treated population compared to placebo population to Week 18 and 20. The NRS endpoint should be recorded weekly (descriptive values), as defined in section 4.2.6 and p-values only provided for the weeks defined in the endpoint.
- Absolute proportion of patients achieving EASI-50 (≥50% improvement from baseline) in treated population compared to placebo population at Week 4, 8, 12, 16, 18 and 20.

- Change from baseline in the Body Surface Area (BSA) affected by AD in treated population compared to placebo population to Week 4, 8, 12, 16, 18 and 20.
- Change from Week 16 in the Body Surface Area (BSA) affected by AD in treated population compared to placebo population to Week 18 and 20.
- Change from baseline in the SCORing Atopic Dermatitis (SCORAD) score in treated population compared to placebo population to Week 4, 8, 12, 16, 18 and 20.
- Change from Week 16 in the SCORing Atopic Dermatitis (SCORAD) score in treated population compared to placebo population to Week 18 and 20.

## 7.4 Efficacy - Exploratory Endpoints Evaluation

All Exploratory efficacy analyses will be performed as described in chapter 6.2 with the FAS only. Change from baseline for exploratory endpoints (vIGA-AD<sup>TM</sup>, SCORAD, DLQI, POEM, AIS and PO-SCORAD) will be analysed using mixed model with repeated measures (MMRM) as described in chapter 7.3.

The following parameters will be analysed as described above:

- Absolut proportion of patients achieving a decrease of at least 2 points in vIGA-AD<sup>TM</sup> in treated population compared to placebo population from baseline to Week 4, 8, 12, 16, 18 and 20.
- Change in proportion of patients achieving a decrease of at least 2 points in vIGA-AD<sup>TM</sup> from Week 16 to Week 18 and 20.
- Change from baseline in the Dermatology Life Quality Index (DLQI) score in treated population compared to placebo population to Week 4, 8, 12, 16, 18 and 20.
- Change from Week 16 in the Dermatology Life Quality Index (DLQI) score in treated population compared to placebo population to Week 18 and 20.
- Change from baseline in the Patient Orientated Eczema Measure (POEM) score in treated population compared to placebo population to Week 4, 8, 12, 16, 18 and 20.
- Change from Week 16 in the Patient Orientated Eczema Measure (POEM) score in treated population compared to placebo population to Week 18 and 20.
- Change in sleep quality assessment (Athens Insomnia Scale) in treated population compared to placebo population from baseline to Week 4, 8, 12, 16, 18 and 20. The AIS endpoint should be recorded weekly (descriptive values), as defined in section 4.2.11 and p-values only provided for the weeks defined in the endpoint.
- Change in sleep quality assessment (Athens Insomnia Scale) in treated population compared to placebo population from Week 16 to Week 18 and 20. The AIS endpoint should be recorded weekly (descriptive values), as defined in section 4.2.11 and p-values only provided for the weeks defined in the endpoint.
- Change from baseline in the Patient-Oriented SCORAD (PO-SCORAD) score in treated population compared to placebo population to Week 4, 8, 12, 16, 18 and 20.
- Change from Week 16 in the Patient-Oriented SCORAD (PO-SCORAD) score in treated population compared to placebo population to Week 18 and 20.

### 7.5 Safety Evaluation

#### **Adverse Events**

The analyses of AEs with onset on or after first administration of study medication ("treatment-emergent AEs") will be conducted with the Safety Analysis Set whereas AEs occurring before first application of study medication will only be listed within the Enrolled Set.

The incidence of AEs will be displayed by MedDRA primary SOC and Preferred Term. The counts in these analyses will reflect numbers of patients reporting one or more AE that map to the MedDRA SOC/preferred term.

For AEs with onset during or after administration of first study medication analysis will be performed for the following AE categories:

- All AEs
- Serious adverse events (SAEs)
- AEs with relationship to the study medication
- AEs leading to discontinuation from study (as documented on the AE page)

Furthermore, a summary table with the overall incidences of the above mentioned AEs will be created.

In addition, the analysis of all treatment emergent AEs will also be done by intensity (mild, moderate and severe) displaying patients who reported more than one intensity for one AE under the worst intensity reported.

Furthermore the analysis of AEs and SAEs will also be done by outcome (Recovered/Resolved, Recovering/Resolving, Not Recovered/Not Resolved, Recovered/Resolved with Sequelae, Fatal and Unknown).

The number/percentage of patients with AEs will also be summarized by MedDRA primary SOC and Preferred Term for most frequent non-serious AEs (incidence of preferred term  $\geq$  5%). In this table, the Totals overall or by SOC will consider only those preferred terms with an incidence >=5%.

All listings will use the Enrolled Set and will include study day of AE onset and AE stop as well as MedDRA information. Note that treatment-emergent AEs are those AEs with an onset at study day 1 or later. Listings will be created for the following topics:

- All AEs
- SAEs
- AEs with relationship to the study medication
- Death (Serious criterion "fatal" or outcome "fatal" documented on the AE page)
- AEs leading to study discontinuation
- AEs before 1st administration of study medication

#### Vital signs

The analysis of vital sign parameters

- Systolic blood pressure [mmHg]
- Diastolic blood pressure [mmHg]
- Heart rate [beats per min]
- Body temperature [°C]
- Body temperature [°F]

will be performed as described in chapter 6.2 with the Safety Analysis Set (descriptive summary of absolute values and changes from baseline).

#### **Physical Examination**

The number and percentage of patients with performed physical examination and the number and percentage of patients with abnormalities during the physical examination will be given within the Safety Analysis Set.

#### **Safety laboratory**

The analyses of the safety laboratory will be performed as described in chapter 6.2 with the Safety Analysis Set. The parameters of clinical chemistry and haematology will be analysed in the standardised units reported by the central laboratory.

In addition the number and percentage of patients with normal values, abnormal values with clinical significance and abnormal values without clinical significance will be given for each parameter of clinical chemistry and haematology. The worst value per patient per study will be used.

Laboratory values outside the normal range will be listed in detail.

Additionally, the change of laboratory values in regard to the respective normal ranges (below, within and above) from baseline to the last value (up to week 26) will be displayed in shift tables for each parameter of clinical chemistry and haematology.

#### ECG data

The analysis of ECG parameters will be performed as described in chapter 6.2 with the Safety Analysis Set. The listing will also include linked AE verbatim(s) and medical history verbatim(s).

#### **Further safety endpoints**

Childbearing Status / Pregnancy test data and virology data will be listed only.

### 7.6 Further Analyses

If not stated otherwise, all further analyses will be performed as described in chapter 6.2 with the Safety Analysis Set.

#### Previous and concomitant medication

The incidence of previous and concomitant medication will be displayed by ATC (Anatomical Therapeutic Chemical) classification (level 1 and 2 and preferred term). The analysis will be performed separately for previous medications and concomitant medications for the Safety Analysis Set. The listing will include a flag indicating if a medication is P (Previous) or C (Concomitant) or PC.

#### **Study medication**

- Duration of intake of study medication [days]
- Number of capsules dispense

will be analysed as described in chapter 6.2 with the Safety Analysis Set.

#### Termination status at end of trial

The incidence and reason for premature study termination (Screening failure, AE, Patient decision (withdrawal of consent to participate), Investigator discretion, Patient lost to follow-up, Lack of efficacy, Pregnancy, Other reasons) will be analysed for the Enrolled Set, i.e. including screening failures and randomised patients, and Safety Analysis Set.

Patients discontinued prematurely will be listed.

The incidence and reason (Violation of Inclusion Criteria X, Violation of Exclusion Criteria Y, Other) for Screening failure will be summarised (using non-randomised subjects of the Enrolled Set only).

#### Study duration and analysis sets

The day of first patient in the study and last patient out of the study will be given for the Enrolled Set as well as for the Safety Analysis Set.

The number of patients in each analysis set will be given by centre and overall. All patients will be listed with their assignment to the analysis populations and if applicable the reason for exclusion from specific analysis sets.

#### Protocol violations

Protocol violations identified in the BDRM will be listed including the decision if these constitute a minor or major protocol violation.

# 8 Tables and Figures

| Item No. | Title | Population | <b>Content Description</b> | Mock<br>Table |
|---|---|---|---|---|
| 14.1.1 | Patient disposition | | | |
| 14.1.1.1 | Patient disposition | Enrolled Set | Descriptive statistics of<br>number of patients in<br>analysis populations by<br>centre and overall | T1 |
| 14.1.1.2 | Study duration | Enrolled Set | Date of first patient in and last patient out | T2 |
| 14.1.1.2.1 | Study duration | SAS | Date of first patient in and last patient out | T2 |
| 14.1.2 | Demographic data | | | |
| 14.1.2.1 | Demographic data I | Randomised<br>Set | Descriptive statistics of continuous variables | Т3 |
| 14.1.2.2 | Demographic data II | Randomised<br>Set | Frequency table of categorical variables | T4 |
| 14.1.3 | Medical history and baseling | e evaluation | | 1 |
| 14.1.3.1 | Medical history /<br>Concomitant diseases by<br>MedDRA primary SOC and<br>preferred term | FAS | Frequency Table | T5 |
| 14.2 | Efficacy | | | |
| 14.2.1 | Primary Endpoint | | | |
| | vIGA-AD <sup>TM</sup> score | | | |
| 14.2.1.1 | vIGA-AD <sup>TM</sup> score by visit | FAS | Frequency table by visit | T4a |
| 14.2.1.2 | vIGA-AD <sup>TM</sup> score by visit and subgroup | FAS | Frequency table by visit and subgroup | T4a |
| 14.2.1.3 | vIGA-AD <sup>TM</sup> response by visit | FAS | Descriptive statistics by visit | T4a |
| 14.2.1.4 | vIGA-AD <sup>TM</sup> response by visit and subgroup | FAS | Descriptive statistics by visit and subgroup | T4a |
| 14.2.1.5 | vIGA-AD <sup>TM</sup> score<br>proportion from baseline to<br>week 16 (GLMM) | FAS | Proportion (n (%) of patients achieving an vIGA-AD <sup>TM</sup> score of 0 (clear) or 1 (almost clear) and a decrease of at least 2 points in vIGA-AD <sup>TM</sup> from baseline to Week 16 using a Generalised Linear Mixed Model | T6.1<br>T6.2 |

| 14.2.1.5.1 | vIGA-AD <sup>TM</sup> score<br>proportion from baseline to<br>week 16 (GLMM) | PPS | Proportion of patients achieving an vIGA-AD <sup>TM</sup> score of 0 (clear) or 1 (almost clear) and a decrease of at least 2 points in vIGA-AD <sup>TM</sup> from baseline to Week 16 using a Generalised Linear Mixed Model | T6.1<br>T6.2 |
|---|---|---|---|---|
| 14.2.1.6 | vIGA-AD <sup>TM</sup> score proportion from baseline to week 16 (GLMM) by subgroup | FAS | Proportion of patients achieving an vIGA-AD <sup>TM</sup> score of 0 (clear) or 1 (almost clear) and a decrease of at least 2 points in vIGA-AD <sup>TM</sup> from baseline to Week 16 using a Generalised Linear Mixed Model by subgroup | T6.1<br>T6.2 |
| 14.2.1.7 | Sensitivity analysis of vIGA-AD <sup>TM</sup> score proportion from baseline to week 16 (de facto estimand) | FAS | Jump to reference method to estimate the de facto estimand | T7.1<br>T7.2 |
| 14.2.1.8 | Sensitivity analysis of vIGA-AD <sup>TM</sup> score proportion from baseline to week 16 (rescue medication) | FAS | Patients who received rescue medication will be evaluated as treatment failures | T6.1<br>T6.2 |
| | EASI-75 score | | | |
| 14.2.1.9 | EASI score by visit | FAS | Descriptive statistics by visit | T3a |
| 14.2.1.10 | EASI score by visit and subgroup | FAS | Descriptive statistics by visit and subgroup | T3a |
| 14.2.1.11 | EASI-75 response by visit | FAS | Descriptive statistics by visit | T4a |
| 14.2.1.12 | EASI-75 response by visit and subgroup | FAS | Descriptive statistics by visit and subgroup | T4a |
| 14.2.1.13 | EASI-75 response from baseline to week 16 (GLMM) | FAS | Proportion of patients<br>achieving EASI-75 (≥75%<br>improvement from<br>baseline) at Week 16 using<br>a Generalised Linear Mixed<br>Model | T6.1<br>T6.2 |

| 14.2.1.13.1 | EASI-75 response from baseline to week 16 (GLMM) | PPS | Proportion of patients<br>achieving EASI-75 (≥75%<br>improvement from<br>baseline) at Week 16 using<br>a Generalised Linear Mixed<br>Model | T6.1<br>T6.2 |
|---|---|---|---|---|
| 14.2.1.14 | EASI-75 response from baseline to week 16 (GLMM) by subgroup | FAS | Proportion of patients<br>achieving EASI-75 (≥75%<br>improvement from<br>baseline) at Week 16 using<br>a Generalised Linear Mixed<br>Model by subgroup | T6.1<br>T6.2 |
| 14.2.1.15 | Sensitivity analysis of<br>EASI-75 response from<br>baseline to week 16 (de<br>facto estimand) | FAS | Jump to reference method to estimate the de facto estimand | T7.1<br>T7.2 |
| 14.2.1.16 | Sensitivity analysis of<br>EASI-75 response from<br>baseline to week 16 (rescue<br>medication) | FAS | Patients who received rescue medication will be evaluated as treatment failures | T6.1<br>T6.2 |
| 14.2.2 | Secondary Endpoints | | , | |
| 14.2.2.1 | vIGA-AD <sup>TM</sup> score | | | |
| 14.2.2.1.1 | vIGA-AD <sup>TM</sup> score<br>proportion from baseline to<br>week 4, 8, 12, 18, 20<br>(GLMM) | FAS | Proportion of patients achieving an vIGA-AD <sup>TM</sup> score of 0 (clear) or 1 (almost clear) and a decrease of at least 2 points in vIGA-AD <sup>TM</sup> from baseline to Week 4, 8, 12, 18 and 20 using a Generalised Linear Mixed Model | T6.1<br>T6.2 |
| 14.2.2.1.2 | Change in vIGA-AD <sup>TM</sup> score proportion at follow-up (GLMM) | FAS | Change in proportion of patients achieving an vIGA-AD <sup>TM</sup> score of 0 (clear) or 1 (almost clear) and a decrease of at least 2 points in vIGA-AD <sup>TM</sup> from Week 16 to Week 18 and 20 using a Generalised Linear Mixed Model | T6.1<br>T6.2 |
| 14.2.2.1.3 | Change in vIGA-AD <sup>TM</sup> | FAS | Change in vIGA-AD <sup>TM</sup> | T8.1 |

| 14.2.2.1.4 | Change in vIGA-AD <sup>TM</sup> score at follow-up (MMRM) | FAS | Change in vIGA-AD <sup>TM</sup> score from week 16 to week 18 and 20 using Mixed Model with Repeated Measures | T8.1<br>T8.2 |
|---|---|---|---|---|
| 14.2.2.1.5 | Change in vIGA-AD <sup>TM</sup> score (mixed ordinal logistic regression) | FAS | Change in vIGA-AD <sup>TM</sup> score using mixed ordinal logistic regression | T9.1<br>T9.2 |
| 14.2.2.2 | EASI score | | | |
| 14.2.2.2.1 | EASI-75 proportion from baseline to week 4, 8, 12, 18, 20 (GLMM) | FAS | Proportion of patients<br>achieving EASI-75 (≥75%<br>improvement from<br>baseline) at Week 4, 8, 12,<br>18 and 20 using a<br>Generalised Linear Mixed<br>Model | T6.1<br>T6.2 |
| 14.2.2.2.2 | Change in EASI score from baseline to week 4, 8, 12, 16, 18, 20 (MMRM) | FAS | Change in EASI score from baseline to week 4, 8, 12, 16, 18, 20 using Mixed Model with Repeated Measures | T8.1<br>T8.2 |
| 14.2.2.2.3 | Change in EASI score at follow-up (MMRM) | FAS | Change in EASI score from week 16 to week 18 and 20 using Mixed Model with Repeated Measures | T8.1<br>T8.2 |
| 14.2.2.2.4 | EASI-50 proportion from baseline to week 4, 8, 12, 16, 18, 20 (MMRM) | FAS | Proportion of patients<br>achieving EASI-50 (≥50%<br>improvement from<br>baseline) at Week 4, 8, 12,<br>18 and 20 | T8.1<br>T8.2 |
| 14.2.2.2.5 | Change in EASI score by visit | FAS | Descriptive statistics by visit | T3a |
| 14.2.2.2.6 | EASI-50 response by visit | FAS | Descriptive statistics by visit | T4a |
| 14.2.2.3 | NRS | 1 | | ı |
| 14.2.2.3.1 | NRS 4 point decrease proportion (MMRM) | FAS | Proportion of patients<br>achieving a decrease of at<br>least 4 points in worst itch<br>NRS from baseline to week<br>4, 8, 12, 16, 18, 20 | T8.1<br>T8.2 |

| 14.2.2.3.2 | NRS 3 point decrease proportion (MMRM) | FAS | Proportion of patients<br>achieving a decrease of at<br>least 3 points in worst itch<br>NRS from baseline to week<br>4, 8, 12, 16, 18, 20 | T8.1<br>T8.2 |
|---|---|---|---|---|
| 14.2.2.3.3 | Change in NRS (MMRM) | FAS | Change from baseline in worst itch NRS to week 4, 8, 12, 16, 18, 20 | T8.1<br>T8.2 |
| 14.2.2.3.4 | Change in NRS at follow-<br>up (MMRM) | FAS | Change from week 16 in worst itch NRS to week 18 and 20 | T8.1<br>T8.2 |
| 14.2.2.3.5 | NRS score by visit | FAS | Descriptive statistics by visit | T3a |
| 14.2.2.3.6 | Change in NRS score | FAS | Descriptive statistics | T3a |
| 14.2.2.3.7 | NRS 3 point decrease and NRS 4 point decrease | FAS | Descriptive statistics | T4a |
| 14.2.2.4 | BSA | | | |
| 14.2.2.4.1 | Change in BSA (MMRM) | FAS | Change from baseline in the body surface area affected by AD to week 4, 8, 12, 16, 18, 20 | T8.1<br>T8.2 |
| 14.2.2.4.2 | Change in BSA at follow-<br>up (MMRM) | FAS | Change from week 16 in<br>the body surface area<br>affected by AD to week 18<br>and 20 | T8.1<br>T8.2 |
| 14.2.2.4.3 | Body Surface Area (Value,<br>Change from Baseline,<br>Change from Wk 16) by<br>visit | FAS | Descriptive statistics of body surface area at baseline and week 4, 8, 12, 16, 18, 20 | ТЗа |
| 14.2.2.5 | SCORAD score | | | |
| 14.2.2.5.1 | Change in SCORAD (MMRM) | FAS | Change from baseline in the SCORAD score to week 4, 8, 12, 16, 18, 20 | T8.1<br>T8.2 |
| 14.2.2.5.2 | Change in SCORAD at follow-up (MMRM) | FAS | Change from week 16 in<br>the SCORAD score to week<br>18 and 20 | T8.1<br>T8.2 |
| 14.2.2.5.3 | SCORAD (Value, Change<br>from Baseline, Change<br>from Wk 16) by visit | FAS | Descriptive statistics by visit | T3a |
| 14.2.2.6 | <b>Exploratory Endpoints</b> | | | |
| | vIGA-AD <sup>TM</sup> score | | | |

| 14.2.2.6.1 | vIGA-AD <sup>TM</sup> score 2 point decrease proportion (MMRM) | FAS | Proportion of patients achieving a decrease of at least 2 points in vIGA-AD <sup>TM</sup> from baseline to Week 4, 8, 12, 16, 18 and 20 | T8.1<br>T8.2 |
|---|---|---|---|---|
| 14.2.2.6.2 | Change in vIGA-AD <sup>TM</sup> score 2 point decrease proportion at follow-up (MMRM) | FAS | Change in proportion of patients achieving a decrease of at least 2 points in vIGA-AD <sup>TM</sup> from Week 16 to Week 18 and 20 | T8.1<br>T8.2 |
| | DLQI score | | | |
| 14.2.2.6.3 | Change in DLQI score (MMRM) | FAS | Change from baseline in the DLQI score to week 4, 8, 12, 16, 18, 20 | T8.1<br>T8.2 |
| 14.2.2.6.4 | Change in DLQI score at follow-up (MMRM) | FAS | Change from week 16 in the DLQI score to week 18 and 20 | T8.1<br>T8.2 |
| 14.2.2.6.5 | DLQI score (Value,<br>Change from Baseline,<br>Change from Wk 16) by<br>visit | FAS | Descriptive statistics by visit | T3a |
| | POEM score | | | |
| 14.2.2.6.6 | Change in POEM score (MMRM) | FAS | Change from baseline in the POEM score to week 4, 8, 12, 16, 18, 20 | T8.1<br>T8.2 |
| 14.2.2.6.7 | Change in POEM score at follow-up (MMRM) | FAS | Change from week 16 in the POEM score to week 18 and 20 | T8.1<br>T8.2 |
| 14.2.2.6.8 | POEM score (Value,<br>Change from Baseline,<br>Change from Wk 16) by<br>visit | FAS | Descriptive statistics by visit | Т3а |
| | <b>Athens Insomnia Scale</b> | | | |
| 14.2.2.6.9 | Change in sleep quality assessment (MMRM) | FAS | Change from baseline in sleep quality assessment (Athens Insomnia Scale) to week 4, 8, 12, 16, 18, 20 | T8.1<br>T8.2 |
| 14.2.2.6.10 | Change in sleep quality assessment at follow-up (MMRM) | FAS | Change from week 16 in sleep quality assessment (Athens Insomnia Scale) to week 18 and 20 | T8.1<br>T8.2 |

| 14.2.2.6.11 | Sleep quality assessment<br>(Value, Change from<br>Baseline, Change from Wk<br>16) by visit | FAS | Descriptive statistics by visit | T3a |
|---|---|---|---|---|
| | PO-SCORAD Score | | | |
| 14.2.2.6.12 | Change in PO-SCORAD score (MMRM) | FAS | Change from baseline in PO-SCORAD score to week 4, 8, 12, 16, 18, 20 | T8.1<br>T8.2 |
| 14.2.2.6.13 | Change in PO-SCORAD score at follow-up (MMRM) | FAS | Change from week 16 in PO-SCORAD score to week 18 and 20 | T8.1<br>T8.2 |
| 14.2.2.6.14 | PO-SCORAD (Value,<br>Change from Baseline,<br>Change from Wk 16) by<br>visit | FAS | Descriptive statistics by visit | T3a |
| 14.2.3 | <b>Further Analyses</b> | | | |
| 14.2.3.1 | Previous medication | SAS | Descriptive statistics by<br>ATC classification (level 1<br>and 2 and preferred term) | T10 |
| 14.2.3.2 | Concomitant medication | SAS | Descriptive statistics by<br>ATC classification (level 1<br>and 2 and preferred term) | T10 |
| 14.2.3.3 | Reason for Termination | Enrolled Set | Frequency Table | T4 |
| 14.2.3.3.1 | Reason for Termination | SAS | Frequency Table | T4 |
| 14.2.3.4 | Screening failure | Non-<br>randomised<br>subjects of<br>the Enrolled<br>Set | Frequency Table | T4 |
| 14.3 | Safety | | | |
| 14.3.1 | Study medication | | | |
| 14.3.1.1 | DS107 intake duration | SAS | Descriptive statistics | T3 |
| 14.3.1.2 | Capsules | SAS | Descriptive statistics of<br>number of capsules<br>dispensed | Т3 |
| 14.3.2 | Adverse events | | | |
| 14.3.2.1 | Summary table of Adverse Events | SAS | Frequency table of patients and number of events per AE category | T11 |
| 14.3.2.2 | Adverse Events by<br>MedDRA SOC and<br>preferred term | SAS | Frequency table | T12 |

| 14.3.2.3 | Serious Adverse Events by<br>MedDRA SOC and<br>preferred term | SAS | Frequency table | T12 |
|---|---|---|---|---|
| 14.3.2.4 | AEs related to DS107 by<br>MedDRA SOC and<br>preferred term | SAS | Frequency table | T12 |
| 14.3.2.5 | AEs leading to study<br>discontinuation by<br>MedDRA SOC and<br>preferred term | SAS | Frequency table | T12 |
| 14.3.2.6 | AEs by SOC, PT and worst intensity | SAS | Frequency table | T13 |
| 14.3.2.7 | AEs by SOC, PT and outcome | SAS | Frequency table | T13 |
| 14.3.2.8 | SAEs by SOC, PT and outcome | SAS | Frequency table | T13 |
| 14.3.2.9 | Most frequent non-serious<br>adverse events by MedDRA<br>SOC and preferred term | SAS | Frequency table | T13 |
| 14.3.5 | Vital signs | | | |
| 14.3.5.1 | Vital signs | SAS | Descriptive Statistics | T3a |
| 14.3.5.2 | Change in vital signs from baseline | SAS | Descriptive Statistics | T3a |
| 14.3.5.3 | ECG | SAS | Descriptive Statistics | T4a |
| 14.3.6 | Laboratory values | | | |
| 14.3.6.1 | Clinical Chemistry & Haematology | SAS | Descriptive Statistics | T3a |
| 14.3.6.2 | Clinical Chemistry &<br>Haematology per category | SAS | Frequency Table (number and percentage of patients with normal values, abnormal values with clinical significance and abnormal values without clinical significance) | T4a |
| 14.3.6.3 | Change in Clinical<br>Chemistry & Haematology | SAS | Shift Table | T14 |
| 14.3.7 | Physical Examination | | | |
| 14.3.7.1 | Physical examination | SAS | Frequency table of patients with physical examination (yes/no) | T4 |

| 14.3.7.2 | Abnormalities during physical examination | SAS | Frequency table of patients with abnormalities during physical examination | Т4 |
|---|---|---|---|---|
| 16 | Appendices | | | |
| 16.2 | Patient data listings | | | |
| 16.2.1 | Patient disposition | Enrolled Set | Individual patient data<br>listing to analysis sets by<br>cohort including reasons for<br>exclusions, if applicable | L1 |
| 16.2.2 | Violations of inclusion/exclusion criteria | Enrolled Set (only patients with violations) | Individual patient data listing by cohort | L6 |
| 16.2.3 | Discontinuation | Enrolled Set | Individual patient data listing including reasons for discontinuation | L2 |
| 16.2.4 | Demographic data /<br>Informed Consent /<br>Randomisation | Randomised<br>Set | Individual patient data listing by cohort | L3 |
| 16.2.5 | Vital Signs | FAS | Individual patient data listing by cohort and visit | L6 |
| 16.2.6.1 | vIGA-AD <sup>TM</sup> score | Enrolled Set | Individual patient data listing by cohort and visit | L6 |
| 16.2.6.2 | EASI score | Enrolled Set | Individual patient data listing by cohort and visit | L6 |
| 16.2.6.3 | NRS score | Enrolled Set | Individual patient data listing by cohort and visit | L6 |
| 16.2.6.4 | BSA | Enrolled Set | Individual patient data listing by cohort and visit | L6 |
| 16.2.6.5 | SCORAD | Enrolled Set | Individual patient data listing by cohort and visit | L6 |
| 16.2.6.6 | DLQI score | Enrolled Set | Individual patient data listing by cohort and visit | L6 |
| 16.2.6.7 | POEM score | Enrolled Set | Individual patient data listing by cohort and visit | L6 |
| 16.2.6.8 | AIS | Enrolled Set | Individual patient data listing by cohort and visit | L6 |
| 16.2.6.9 | PO-SCORAD score | Enrolled Set | Individual patient data listing by cohort and visit | L6 |

| 16.2.7 | <b>Adverse Events Listings</b> | | | |
|---|---|---|---|---|
| 16.2.7.1 | Adverse events | Enrolled Set | Individual patient data listing by cohort | L4 |
| 16.2.7.2 | Serious adverse events | Enrolled Set | Individual patient data listing by cohort | L4 |
| 16.2.7.3 | AEs related to DS107 | Enrolled Set | Individual patient data listing by cohort | L4 |
| 16.2.7.4 | AEs leading to death | Enrolled Set | Individual patient data listing by cohort | L4 |
| 16.2.7.5 | AEs leading to study discontinuation | Enrolled Set | Individual patient data listing by cohort | L4 |
| 16.2.7.6 | AEs before first administration of DS107 | Enrolled Set | Individual patient data listing by cohort | L4 |
| 16.2.8 | Listing of individual laboratory measurements | | | |
| 16.2.8.1 | Laboratory values | SAS | Individual patient data<br>listing of laboratory results<br>(haematology, clinical<br>chemistry) | L5 |
| 16.2.8.2 | Laboratory values outside the normal range | SAS | Individual patient data listing of laboratory results outside the normal range | L5 |
| 16.2.9 | Other Listing | | | |
| 16.2.9.1 | Physical examinations | SAS | Individual patient data listing by cohort and visit | L6 |
| 16.2.9.2 | Medical History /<br>Concomitant diseases | FAS | Individual patient data listing by cohort | L6 |
| 16.2.9.3 | Childbearing status and<br>Pregnancy test data | FAS | Individual patient data listing by cohort and visit | L6 |
| 16.2.9.4 | Virology | FAS | Individual patient data listing by cohort | L6 |
| 16.2.9.5 | ECG | FAS | Individual patient data listing by cohort and visit | L6 |
| 16.2.9.6 | Study drug dispensed | SAS | Individual patient data listing by cohort and visit | L6 |
| 16.2.9.7 | Patient diary compliance | SAS | Individual patient data listing by cohort and visit | L6 |
| 16.2.9.8 | IMP accountability and IMP compliance | SAS | Individual patient data listing by cohort and visit | L6 |
| 16.2.9.9 | Previous and Concomitant medication | FAS | Individual patient data listing by cohort | L6 |

## Statistical Analysis Plan DS107G-05-AD3 Version 1.0 (final), 24-Sep-2020

| 16.2.9.10 | Violations of inclusion/exclusion criteria | Enrolled Set<br>(only<br>patients with<br>violations) | Individual patient data listing by cohort | L6 |
|---|---|---|---|---|
| 16.2.9.11 | Protocol violations | SAS | Individual patient data listing by cohort | L6 |

#### 9 References

- Carpenter, JR, Roger, JH & Kenward, MG 2013. 'Analysis of longitudinal trials with protocol deviations: a framework for relevant, accessible assumptions, and inference via multiple imputation.' *J Biopharm Stat*; 23(6), pp. 1352-71.
- Hanifin, JM, Thurston, M, Omoto, M, Cherill, R, Tofte, SJ, & Graeber, M 2001.
   'The eczema area and severity index (EASI): assessment of reliability in atopic dermatitis. EASI Evaluator Group.' Exp Dermatol. Feb;10(1), pp. 11-8.
- Phan, NQ, Blome, C, Fritz, F, Gerss, J, Reich, A, Ebata, T, Augustin, M, Szepietowski, JC & Ständer, S 2012. 'Assessment of pruritus intensity: prospective study on validity and reliability of the visual analogue scale, numerical rating scale and verbal rating scale in 471 patients with chronic pruritus.' Acta Derm Venereol; 92 pp. 502–507.
- Soldatos CR, Dikeos DG, Paparrigopoulos TJ: Athens Insomnia Scale: validation of an instrument based on ICD-10 criteria. Journal of Psychosomatical Research 48 (2000) 555-560.